CLINICAL TRIAL: NCT01735825
Title: Prospective Randomised Study Comparing Efficacy of Treatment Coronary In-stent Restenosis Using Drug Eluting Paclitaxel-coated Balloon and Drug Eluting Stent With Everolimus.
Brief Title: Treatment of Coronary In-Stent Restenosis
Acronym: TIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNO-KVO 631/2011 Pleva
Record Dates: First submitted 2012-11-07; First posted 2012-11-28 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Restenosis
Keywords: coronary artery disease; stent; restenosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Intervention Model Description: iopromide coated paclitaxel-eluting balloon catheter
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- iopromide paclitaxel-eluting balloon (Experimental): Patients with coronary in-stent restenosis treated by drug eluting paclitaxel-coated balloon catheter (iopomide coating)
  Interventions: Device: paclitaxel-coated balloon catheter with Iopromide coating
- drug eluting stent (Active Comparator): Patients with coronary in-stent restenosis treated by drug eluting stent with everolimus
  Interventions: Device: drug eluting stent with everolimus
- seal-wing PEB (Other): Observational, non-randomised arm:
  Pts with ISR treated by seal-wing paclitaxel-eluting balloon catheter
  Interventions: Device: seal-wing paclitaxel-eluting balloon catheter

INTERVENTIONS:
Device: paclitaxel-coated balloon catheter with Iopromide coating — Patients with coronary in-stent restenosis treated by drug eluting paclitaxel-coated balloon catheter
  Other Names: Sequent Please
  Arms: iopromide paclitaxel-eluting balloon
Device: drug eluting stent with everolimus — Patients with coronary in-stent restenosis treated by drug eluting stent with everolimus
  Other Names: Promus
  Arms: drug eluting stent
Device: seal-wing paclitaxel-eluting balloon catheter — Patients with coronary in-stent restenosis treated by seal-wing paclitaxel-eluting balloon catheter
  Other Names: Protege
  Arms: seal-wing PEB

SUMMARY:
The purpose of this study is to compare efficacy of coronary in-stent restenosis therapy using drug eluting paclitaxel-coated balloon catheters with the latest generation of drug eluting stents releasing everolimus.

DETAILED DESCRIPTION:
In-stent restenosis after coronary angioplasty is currently one of the main limitations of this method, leading to a recurrence of exertional angina pectoris or manifesting as acute coronary syndrome. Histopathologic substrate of in-stent restenosis is neointimal hyperplasia.

Repeated plain balloon angioplasty or using cutting balloon catheters in the treatment of in-stent restenosis does not achieve satisfactory results. Brachytherapy, used in the past, it has also abandoned. The current treatment of in-stent restenosis is the use of drug eluting stents. Local drug released from these stents prevents new neointimal hyperplasia.This treatment carries the risk of late thrombosis (due to delayed neoendotelization) the stent struts and requires rigorous long-term dual antiplatelet therapy with the risk of bleeding complications. The drug-coated balloon catheters provide short-term penetration of the active substance into the vascular wall, leading to the inhibition of hyperproliferation vascular smooth muscle cells, but due to short-term effect they do not affect negatively stent struts neoendotelization. Comparable effects of in-stent restenosis therapy using paclitaxel releasing balloons was demonstrated in comparison with paclitaxel releasing stents, however, the development of drug eluting stents meanwhile progressed. The aim of our study is to compare efficacy of coronary in-stent restenosis therapy using drug eluting paclitaxel-coated balloon catheters with the latest generation of drug eluting stents releasing everolimus. Primary endpoint of our study is late lumen loss, because it represents accurate angiographic parameter predicting the need for repeat revascularisation and thus the clinical benefit for the patient.

The 3rd observational, non-randomised arm compares the treatment with seal-wing paclitaxel-eluting balloon with two randomised arms (PEB vs. EES).

3-year long term clinical follow-up of iopromide-coated PEB and EES arms was performed. All clinical MACE (CV death, AMI and TVR) were recorded.

Subanalysis of seal-wing PEB arm comparrng the treatment of BMS and DES-ISR was added.

ELIGIBILITY:
Inclusion Criteria:

* history of percutaneous coronary intervention with stent placement
* verified coronary in-stent restenosis suitable for percutaneous re-intervention
* signed informed consent

Exclusion Criteria:

* contraindication to long term dual antiplatelet therapy
* increased risk of bleeding
* known generalized malignancy
* pregnancy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Late lumen loss | 12 month
  Late loss was defined as the minimal vessel lumen diameter immediately after the procedure minus the lumen diameter at angiographic follow-up

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 12 month
  Major Adverse Cardiac Events are defined as cardiovascular death, acute myocardial infarction or target vessel revascularisation

OTHER OUTCOMES:
Binary restenosis | 12 month
  Binary restenosis is defined as a > 50% diameter stenosis at angiographic follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Leos Pleva, M.D., Principal Investigator — Cardiovascular Department, University Hospital Ostrava, Czech Republic
Locations (1):
- University Hospital, Ostrava, Czechia

REFERENCES:
- [Background] 1.TAXUS III Trial: In-Stent Restenosis Treated With Stent-Based Delivery of Paclitaxel Incorporated in a Slow-Release Polymer Formulation J. van der Giessen, Circulation 2003,107:559-564: 2.Sirolimus-eluting stent or paclitaxel-eluting stent vs balloon angioplasty for prevention of recurrences in patients with coronary in-stent restenosis: a randomized controlled trial. Kastrati A,JAMA 2005;293:165-71 3.Treatment of coronary in-stent restenosis with a paclitaxel-coated ballon catheter, B.Scheller, NEJM,355;20,Nov 16,2006 4.Randomized Trial of Paclitaxel- Versus Sirolimus-Eluting Stents for Treatment of Coronary Restenosis in Sirolimus-Eluting Stents The ISAR-DESIRE 2 Study. Mehilli J, J Am Coll Cardiol 2010 Mar 5 5.Everolimus-eluting versus paclitaxel-eluting stents in coronary artery disease. Stone GW,. N Engl J Med 2010 May 6;362:1663-74 6.Angiogaphic surrogate end points in drug-eluting stent trials, S.J.Pocock, JACC, Vol 51,No 1,2008
- [Derived] Pleva L, Kukla P, Zapletalova J, Hlinomaz O. Long-term outcomes after treatment of bare-metal stent restenosis with paclitaxel-coated balloon catheters or everolimus-eluting stents: 3-year follow-up of the TIS clinical study. Catheter Cardiovasc Interv. 2018 Nov 15;92(6):E416-E424. doi: 10.1002/ccd.27688. Epub 2018 Jul 18. PMID 30019843
- [Derived] Pleva L, Kukla P, Zapletalova J, Hlinomaz O. Efficacy of a seal-wing paclitaxel-eluting balloon catheters in the treatment of bare metal stent restenosis. BMC Cardiovasc Disord. 2017 Jun 26;17(1):168. doi: 10.1186/s12872-017-0602-6. PMID 28651572
- [Derived] Pleva L, Kukla P, Kusnierova P, Zapletalova J, Hlinomaz O. Comparison of the Efficacy of Paclitaxel-Eluting Balloon Catheters and Everolimus-Eluting Stents in the Treatment of Coronary In-Stent Restenosis: The Treatment of In-Stent Restenosis Study. Circ Cardiovasc Interv. 2016 Apr;9(4):e003316. doi: 10.1161/CIRCINTERVENTIONS.115.003316. PMID 27069104